CLINICAL TRIAL: NCT04377321
Title: Colchicine Has Anti-diabetic Effect and May be an Option for Type 2 Diabetes Management
Brief Title: Colchicine Has Anti-diabetic Effect
Status: Completed | Type: Observational
Sponsor: Ministry of Health and Population, Egypt (Other Government)
Responsible Party: Principal Investigator, mahmoud younis, consultant, Ministry of Health and Population, Egypt
Other Study IDs: ymodmenna@gmail.com
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Treatment Adherence
Keywords: type 2 diabetes; colchicine; inflammatory markers
MeSH Terms: conditions — Treatment Adherence and Compliance; Diabetes Mellitus, Type 2 | interventions — Colchicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- group 1 on cochicine: The first group patients received colchicine 0.5 twice daily for 6 months
  Interventions: Drug: Colchicine Tablets
- group 2 on glucophage 1 gm twice daily: second group received glucophage 1gm twice daily for 6 months
  Interventions: Drug: Colchicine Tablets
- group 3 control: the third group patients were on diet only for 6 months
  Interventions: Drug: Colchicine Tablets

INTERVENTIONS:
Drug: Colchicine Tablets — colchicine tabletes for 6 months

SUMMARY:
Colchicine has antidiabetic effect and may be an option for type 2 diabetes management

DETAILED DESCRIPTION:
Observational cohort prospective study with following of 150 newly diagnosed type 2 diabetes patients who were in 3 groups, had been monitored in a private clinic, each group 50 patients number, with 30 females and 20 males after written consent from all patients. The ages of all patients were between 35 and 55 years.

The aim of this study was to evaluate colchicine effect on A1C of newly diagnosed type2 diabetes compared to the metformin and control group on diet only.

The first group patients received colchicine 0.5twice daily for 6 months, the second group received metformin 1gm twice daily, the third group patients were on diet only. During the period of treatment, the investigators followed the patients if there were side effects of the drugs used. No side effects were monitored during the period of treatment except for gastric upset in some patients using metformin

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes newly diagnosed age 35- 55 years

Exclusion Criteria:

* severe anemia hypothyroidism and hyperthyroidism moderate to severe liver or kidney disease

Ages: 35 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Observational cohort prospective study with following of 150 newly diagnosed type 2 diabetes patients who were in 3 groups, had been monitored in a private clinic, each group 50 patients number, with 30 females and 20 males after written consent from all patients. The ages of all patients were between 35 and 55 years.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
colchicine for treatment of type diabetes patients | 6 months
  colchicine tablets .5 mg twice daily for 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud Younis, Cairo, Egypt